CLINICAL TRIAL: NCT00714194
Title: The Effect of Daily Interruption of Continuous Sedation on the Occurrence of Delirium and Perception of Sleep in ICU Patients
Brief Title: Effect of Daily Interruption of Continuous Sedation on Delirium, Sleep Perception in Intensive Care Unit (ICU) Patients
Acronym: ICUDelirium
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H41297-32404-01
Record Dates: First submitted 2008-06-16; First posted 2008-07-14 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Delirium; Sleep Perception
Keywords: sedation; delirium; sleep; sedation withdrawal; ICU patients
MeSH Terms: conditions — Delirium | interventions — Lorazepam; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Patients in the control group will receive continuous sedative infusions without daily interruption of sedatives based on the standard clinical practice of the TICU.
  Interventions: Procedure: Normal continuous sedation
- 2 (Experimental): Patients in the intervention group will receive daily interruption of sedative.
  Interventions: Other: Daily interruption of continuous sedation

INTERVENTIONS:
Procedure: Normal continuous sedation — Normal continuous sedation.
  Arms: 1
Other: Daily interruption of continuous sedation — Withdrawal of normal continuous sedation with Lorazepam, Midazolam, and Propofol from 7:00 am to 8:00 am daily until continuous sedation discontinuation.
  Other Names: Ativan®, Versed®, Driprivan®
  Arms: 2

SUMMARY:
This is an intervention study whose purpose is to determine whether daily interruption of sedative infusion contributes to the reduction of the occurrence of delirium and improves sleep perception in critically ill patients. Patients in a trauma intensive care unit (TICU) receiving mechanical ventilation and continuous infusion of sedatives will be enrolled in the study. A patient will be entered into the study after the family member has consented to have the patient participate.

DETAILED DESCRIPTION:
This is an intervention study whose purpose is to determine whether daily interruption of sedative infusion contributes to the reduction of the occurrence of delirium and improves sleep perception in critically ill patients. Patients in a trauma intensive care unit (TICU) receiving mechanical ventilation and continuous infusion of sedatives will be enrolled in the study. A patient will be entered into the study after the family member has consented to have the patient participate. A sequential assignment method will be used to compare two groups of 20 patients in each group. The first group of 20 patients (control group [CG]) to be studied will receive continuous sedative infusion without daily interruption. The second group of 20 patients (intervention group [IG]) will receive a daily interruption of sedative infusion.

If control and intervention group data are not sufficient to elicit the effect of daily interruption of sedatives, data collection will continue using the sequential assignment method alternating control and intervention group 10 patients at a time. This method will proceed until an effect is detected or until the a priori sample size of 182 (i.e., 91 patients per group) has been reached.

The intervention group will be monitored during the daily interruption of sedative infusion (i.e., sedation wake-up trial[SWT])in order to measure the following variables: delirium, physiological response (heart rate [HR], respiratory rate [RR], blood pressure [BP], and pulse oxygen saturation [SpO2]), pain intensity, and agitation/sedation level.Once the patient is awake during the SWT period, the patient will be screened for SBT. If the patient meets the SBT criteria, then the mechanical ventilator mode will be changed to continuous positive airway pressure (CPAP) or the patient will be placed in a T-tube circuit for 2 hours or until the patient presents signs of SBT failure. Delirium will be measured 3 times a day for a maximum of 3 days in both groups after continuous deep sedation discontinuation using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Sleep perception will be measured by a sleep questionnaire (Sleep Perception in the ICU) after discontinuous of continuous sedation. Agitation/sedation level will be measured with the Richmond Agitation-Sedation Scale (RASS) and Bispectral Index (BIS), and pain intensity with a 0 to 10 numeric rating scale (NRS).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 21 years will be recruited from a Trauma Intensive Care Unit of Puerto Rico. This unit receives critically ill patients with three or more affected body systems involved after motor vehicle accident, gunshot injury, penetrating injury, and falls.

Exclusion Criteria:

* Baseline neurological diseases
* Head trauma or acute neurological injury with Glasgow Coma Scale score < 8
* Death expected within 24 hours (APACHE II ≥ 30)
* History of alcoholism
* History of drug dependence
* Deaf and blind patients

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Delirium and sleep | 3 days in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine V Padilla, PhD, Study Chair — The Regents of the University of California, San Francisco
Locations (1):
- Trauma Unit University of Puerto Rico Medical Center, San Juan, Puerto Rico